CLINICAL TRIAL: NCT01577212
Title: Individualized Dose Escalation for Non-small Cell Lung Cancer (NSCLC) Using Volumetric Modulated Arc Therapy (VMAT)
Brief Title: Individualized Dose Prescription in Advanced Stage Lung Cancer Patients Using Modern (Chemo)Radiotherapy
Acronym: IDEAL-VMAT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Jan Bussink, Associate Professor, Radboud University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMO 2011/345; NL nr 35536.091.11 (Registry Identifier: CCMO)
Record Dates: First submitted 2012-03-16; First posted 2012-04-13 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Stage III Non-small Cell Lung Cancer; Individualized Radiation Dose Escalation
Keywords: stage III NSCLC; (chemo)radiotherapy; individualized dose-escalation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Individualized dose escalation (Experimental): Individualized dose escalation on the basis of the dose to the organs at risk.
  Interventions: Radiation: Individualized dose escalation

INTERVENTIONS:
Radiation: Individualized dose escalation — Individualized dose escalation on the basis of the maximally tolerable dose to organs at risk - lung, esophagus, spinal cord, heart, brachial plexus

SUMMARY:
The aim of this present study is to test the feasibility and toxicity of individualized hypofractionated radiotherapy, and to report outcome data. In case this phase II trial has favorable results, a phase II/III trial on maximally tolerable, individualized, hypofractionated radiotherapy within a shorter overall-treatment time is aimed for.

DETAILED DESCRIPTION:
In the Netherlands, approximately 10.000 new patients are diagnosed with lung cancer every year. Of these, 80% present with non-small-cell lung cancer. Between 1995 and 2008, the national incidence has risen with 16% caused by an impressive increase of 53% in women suffering from this disease. The aggressive nature of this disease leads to a one-year survival rate of 45% and a 5-year survival rate of only 14%.

It is widely accepted that surgery provides the best chance of cure in patients with operable NSCLC (www.oncoline.nl). In practice, only 20% of patients are amenable for tumor resection with curative intent. Alternatively, stereotactic body radiation therapy (SBRT) results in excellent local control in localized early stage disease.

In locally advanced, inoperable disease, combined chemotherapy and external-beam radiotherapy (EBRT) are increasingly being used. Evidence suggests that concurrent schedules are more effective than sequential treatments despite increased toxicity, although the true magnitude of the additional benefit remains uncertain. However, a large number of patients with locally advanced NSCLC is not suitable for concurrent chemoradiotherapy due to their general condition, age, comorbidity or tumor-related factors. Therefore, there is a need to increase effectiveness of treatment for all patients with advanced stage NSCLC undergoing either radiotherapy alone, neoadjuvant chemotherapy followed by radiotherapy, or concurrent treatment.

Apart from the addition of chemotherapy, treatment modification by intensification of the radiotherapy schedule or by dose escalation has been proven beneficial. Several phase I/II trials explored altered EBRT fractionation schedules that increased the biological effective dose to the primary tumor and reduced local relapse rate. Thereby, two main principles were pursued: reduction of the dose per fraction (≤ 1.8 Gy), giving two or three fractions per day (so-called hyperfractionation), aimed at sparing normal tissues while increasing the dose to the primary tumor; increase of the fraction dose (≥ 2 Gy), combined with a reduction in the total number of fractions (so-called hypofractionation) aimed at increasing the effective tumor dose in less radiation-sensitive primary tumors. On the one hand, hyperfractionation limits the treatment-related side-effects, on the other hypofractionation is attractive for the patient and radiation department as the number of treatment fractions can be reduced.

Intensification of the irradiation schedule by continuous, hyperfractionated radiotherapy (CHART) delivered in 12 consecutive days showed an absolute improvement in two-year survival. With the advent of highly conformal dose planning and delivery techniques during the last decade (i.e., 3-dimensional conformal radiation therapy, 3D-CRT; intensity-modulated radiation therapy, IMRT; volumetric-modulated arc therapy, VMAT/RapidArc; Tomotherapy), organ-sparing technology became widely available. Recently, van Baardwijk and collaborators published an individualized dose prescription study in 166 stage-III NSCLC patients. Already in 2006, Belderbos et al. reported favorable toxicity data and an encouraging failure-free interval in 88 inoperable NSCLC patients treated with intensified, hypofractionated 3D-CRT based on the MTD to the lung.

Apart from these reported studies, there are three hypofractionation trials being conducted elsewhere. In the UK, two 3D-CRT based phase I/II trials have been approved investigating individualized dose escalation based on normal tissue dose constraints in patients with stage II or stage III NSCLC (ISRCTN12155469 and I-START; CRUK/10/005). In the US, the University of Wisconsin is conducting a helical tomotherapy-based hypofractionation study (NCT00214123) with pulmonary toxicity (pneumonitis grade 3 lasting for more than 2 weeks) as primary endpoint.

The reported hypo- and hyperfractionation studies have a 'trial-and-error' approach for dose-level estimation in common. In a recent in silico trial in 26 stage III NSCLC patients, we have investigated the use of a dedicated software tool for individual dose escalation by hypofractionation. Based on an existing, clinical IMRT/VMAT treatment plan (66 Gy in 33 fractions), radiation dose was escalated by scaling the radiation dose until the maximum tolerated dose constraints for the healthy lung, the esophagus, spinal cord, brachial plexus or heart was met. The aim of this present study is to test the feasibility and toxicity of individualized hypofractionated radiotherapy, and to report outcome data. In case this phase II trial has favorable results, a phase II/III trial on maximally tolerable, individualized, hypofractionated radiotherapy within a shorter overall-treatment time is aimed for.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed stage IIIA/B NSCLC (excluding pleural effusion and mixed pathology)
2. Irresectable disease (as assessed by multidisciplinary team) or patient refusing surgery
3. Disease which can be encompassed within a radical radiotherapy treatment plan in keeping with standard practice at the participating center
4. Proposed treatment consists of radiotherapy alone or concurrent chemoradiation
5. WHO performance status 0 or 1
6. Adequate respiratory function: FEV1 ≥ 1.5 L and DLCO > 40%, predicted on baseline pulmonary function tests
7. Age ≥ 18 years, no upper age limit
8. Estimated life expectancy of more than 6 months
9. Patient is available for follow-up
10. Written informed consent obtained

Exclusion Criteria:

1. Clinically diagnosed NSCLC
2. Previous or current malignant disease likely to interfere with the protocol treatment or comparisons
3. Prior thoracic radiotherapy
4. Proposed treatment consist of sequential chemoradiation
5. Prior lobectomy / pneumonectomy
6. Prior chemotherapy using gemcitabine or bleomycine
7. Superior sulcus tumors if the brachial plexus is within the high-dose volume
8. Medically unstable (e.g., ischaemic heart disease, esophageal disorders)
9. Pregnancy
10. Connective tissue disorders
11. Abnormal kidney function interfering with administration of iv contrast agent (GFR<60)
12. Uncontrolled diabetes mellitus hampering 18FDG-PET
13. Inability to comply with protocol or trial procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pulmonary toxicity grade 2-4 | 2 years
Esophageal toxicity grade 2-4 | 2 years

SECONDARY OUTCOMES:
Increase in tumor control probability (TCP) | 2 years
Local-regional failure | 2 years
Progression-free survival | 2 years
Quality of life | 2 years
Overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan Bussink, MD PhD, Principal Investigator — Radboud University Medical Center; Esther GC Troost, MD PhD, Principal Investigator — Radboud University Medical Center; Robin Wijsman, MD, Principal Investigator — Radboud University Medical Center; Aswin L Hoffmann, MSc, Principal Investigator — Maastro Clinic, The Netherlands; Lioe-Fee de Geus-Oei, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands